CLINICAL TRIAL: NCT02660398
Title: Incidence and Severity of Residual Neuromuscular Blockade With Application of a Protocol for Paralysis and Neostigmine Reversal of Rocuronium
Brief Title: Incidence and Severity of Residual Neuromuscular Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Stephan Thilen, Assistant Professor, Anesthesiology, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 50608
Record Dates: First submitted 2016-01-15; First posted 2016-01-21 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Residual Neuromuscular Blockade
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controls (No Intervention): Our control group will consist of an observational cohort of 40 patients in whom we will make quantitative assessments of the Train-of-four ratio (TOF ratio). This is done using the TOF-Watch SX monitor. The monitor will be calibrated after induction of general anesthesia, measurement of the TOF ratio will be obtained at time of extubation and again at the time of arrival to the Post Anesthesia Care Unit (PACU).
- Intervention (Other): The intervention consists of a protocol for intraoperative management of neuromuscular blockade with rocuronium and reversal with neostigmine. A train-of-four count of 4 at the thumb will be confirmed prior to administration of an adjusted dose of neostigmine. TOF ratio is measured in the same manner as for the Control group, it is done using the TOF-Watch SX monitor. The monitor will be calibrated after induction of general anesthesia, measurement of the TOF ratio will be obtained at time of extubation and again at the time of arrival to the Post Anesthesia Care Unit (PACU).
  Interventions: Procedure: Standardized NMBD Management

INTERVENTIONS:
Procedure: Standardized NMBD Management — The intervention phase will introduce a standardized research protocol that spells out NMBD management, including how muscle relaxant should be administered and monitored, and how reversal with neostigmine should be done.
  Arms: Intervention

SUMMARY:
This prospective study will take place at Harborview Medical Center (HMC) and the University of Washington Medical Center (UWMC), and will enroll adult patients undergoing abdominal surgery. The purpose of this study is to identify if the use of a specific plan to managing muscle relaxants will help decrease the risk of muscle weakness after general anesthesia with muscle relaxation in a population of patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
80 patients will be enrolled in this prospective study. The first 40 patients will serve as controls and will not have an intervention.

Patients who have surgery and receive general anesthesia often receive muscle relaxants called neuromuscular blocking drugs or NMBDs. NMBDs facilitate anesthesiologists' performance of tracheal intubation, provide muscle relaxation during surgery, and are sometimes administered to prevent movement. After surgery, an anesthesiologist monitors how the muscle relaxants wear off, and gives a drug to help reverse the effect of the NMBDs before the tracheal breathing tube is removed and a patient is awakened and taken to the postoperative care area (PACU).

A patient who receives NMBDs for their routine care can experience a leftover effect of the drug after their general anesthesia wears off. This condition is called Residual Neuromuscular Blockade. The management of NMBDs in patients for routine care vary by anesthesia provider. This study will explore if the use of a specific plan to managing muscle relaxants will help decrease the risk of muscle weakness after general anesthesia. Anesthesiologists routinely use peripheral nerve stimulators to assess the degree of muscle relaxation. Very commonly a series of 4 electrical stimulations are given over 2 seconds and each stimulation result in a twitch of the thumb when the ulnar nerve is stimulated at the wrist. This is called train-of-four (TOF) monitoring. When the patient is deeply relaxed, then all twitches are not present but as the drug effect diminishes over time, the twitches return. When 4 twitches are present, an exact measurement of the so-called TOF ratio can be calculated if an objective monitor is used. The ratio is the strength of the fourth twitch divided by the strength of the first twitch. The most commonly used reversal drug is neostigmine and it is known from previous research that it works more effectively if the muscle relaxation is not profound. In the intervention group, the investigators will confirm that the neuromuscular blockade has spontaneously recovered to a level where all 4 thumb twitches are present before neostigmine is administered.

All patients will have objective measurements obtained using the FDA approved monitor TOF-Watch SX. This monitor will be applied at the beginning of each case and will be calibrated immediately after induction of anesthesia. This is a simple automated process that takes less than 1 minute. The investigators will also obtain a TOF ratio measurement at the beginning of the case, before a muscle relaxant has been administered. This initial measurement allows for normalization of postoperative measurements. Measurement will be obtained again at the time of extubation, i.e. the removal of the breathing tube, which usually occurs in the operating room as the patient is awakened after surgery. Patients are routinely transferred to the post-anesthesia care unit (PACU) within minutes of being extubated and shortly after arrival to the PACU, the anesthesiologists transfers the care to PACU RNs. The investigators will obtain one more TOF-ratio measurement when the patient has just arrived to the post-anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older
* Will undergo open or laparoscopic abdominal surgery expected to last <6 hours at HMC or UWMC
* Have ASA physical status I-III
* Scheduled to have general anesthesia with at least 1 dose of nondepolarizing NMBD for endotracheal intubation or maintenance of neuromuscular block (NMB)

Exclusion Criteria:

* Allergy to NMBDs
* Patients with neuromuscular disease (myasthenia gravis or muscular dystrophy)
* Pregnant or lactating women
* Non-English speaking
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of residual paralysis | The outcome measure will be assessed at time of extubation
  The incidence of residual paralysis defined as a TOF ratio <0.9 will be measured.

SECONDARY OUTCOMES:
Incidence of severe residual paralysis | The outcome measure will be assessed at time of extubation
  The incidence of severe residual paralysis defined as a TOF ratio <0.7 will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Thilen, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thilen SR, Ng IC, Cain KC, Treggiari MM, Bhananker SM. Management of rocuronium neuromuscular block using a protocol for qualitative monitoring and reversal with neostigmine. Br J Anaesth. 2018 Aug;121(2):367-377. doi: 10.1016/j.bja.2018.03.029. Epub 2018 May 19. PMID 30032875